CLINICAL TRIAL: NCT00553436
Title: Evaluation of an Endoscopic Suturing System for Tissue Apposition in Colonic Polypectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Amy Mahanes, Ethicon Endo-Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-07-0004; UH IRB #07-07-08
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2010-03-26 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Polyps
Keywords: colon; rectum; polyp; EMR; Established indication for a procedure greater than colonoscopy and colonic polypectomy
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enrolled Subjects treated with TAS device (Experimental): All enrolled subjects treated with the Tissue Apposition System (TAS) device
  Interventions: Device: Tissue Apposition System (TAS) Device

INTERVENTIONS:
Device: Tissue Apposition System (TAS) Device — Closure of defect following polypectomy using the Tissue Apposition System (TAS) Device.

SUMMARY:
The purpose of this study is to show that the surgical site in the bowel wall can be sewn closed in the colon or intestine, with a new sewing device after removal of a benign polyp according to standard of care.

DETAILED DESCRIPTION:
Polypectomy is the medical term for removing polyps. Polyps are abnormal like growths that protrude into the lining of the bowel. Because a polyp cannot always be removed by a snare, the usual and simplest method, (for example, it may be too flat), a doctor (colorectal surgeon) may perform a polypectomy using a technique called Endoscopic Mucosal Resection (EMR). Endoscopic Mucosal Resection (EMR)is based on the concept that endoscopy (looking at the inside of your colon with an instrument called a colonoscope) provides visualization and access to the innermost lining of the gastrointestinal tract, where a polyp originates. The Endoscopic Mucosal Resection (EMR)performed during this study will be standard of care according to the current practice at University Hospitals of Cleveland.

Following polyp removal, the study procedure will be performed. A medical device is being evaluated to help with this procedure by closing the wound that remains after the polyp is removed without performing an open surgical operation. This involves suturing (sewing) the tissue back together with a Tissue Apposition System (TAS). This is also called tissue approximation. The sewing device being evaluated has been cleared by the Food and Drug Administration (FDA).

Up to 20 men and women, at least 21 years of age, requiring removal of a colonic or rectal polyp that cannot be removed by traditional colonic polypectomy, will be asked to enroll in the study. Following polyp removal, these patients will have the remaining tissue area closed using the study sewing device. Participation in this study will last approximately three months.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age;
* Willing to give consent and comply with evaluation and treatment schedule;
* Approved for polypectomy per standard preoperative endoscopic evaluation;
* Established indication for a procedure greater than colonoscopy and colonic polypectomy. This will include polyps not suitable for current practice (snare procedure) endoscopic resection by nature of size or location, in which an intestinal resection, laparoscopic-assisted polypectomy is required;
* Surgical area viewable with laparoscopy.

Exclusion Criteria:

* Physical or psychological condition which would impair study participation;
* Unable or unwilling to attend follow-up visits and examinations;
* Concurrent surgical procedure;
* Pregnancy;
* A polyp which appears to be an invasive cancer, even with negative pathology;
* A polyp with biopsies suspicious for invasive cancer;
* Participation in any other investigational device or drug study within 30 days prior to enrollment; or
* Any condition which precludes compliance with the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Conor P Delaney, MD MCh PhD FRCSI FACS, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Agrawal D, Chak A, Champagne BJ, Marks JM, Delaney CP. Endoscopic mucosal resection with full-thickness closure for difficult polyps: a prospective clinical trial. Gastrointest Endosc. 2010 May;71(6):1082-8. doi: 10.1016/j.gie.2009.12.036. PMID 20438900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single Center, hospital based surgical suite. Enrollment from 20 August 2007 to 09 April 2009.
Pre-assignment Details: Non-randomized. Patients were considered for enrollment based on inclusion / exclusion criteria and were offered the opportunity for enrollment. Those that signed informed consent were enrolled.
Groups:
- Enrolled Subjects Treated With Tissue Apposition System (TAS): All enrolled subjects treated with Tissue Apposition System (TAS) device and achieving defect closure
Period: Overall Study
Arm/Group | Enrolled Subjects Treated With Tissue Apposition System (TAS)
Started | 7 (20 August 2007)
Completed | 6 (09 April 2009)
Not Completed | 1
Not completed — Conversion to another procedure | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enrolled Subjects Treated With Tissue Apposition System (TAS)
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Secondary Outcome: Numbers of Participants With Successful Deployments of Tissue Anchors and Associated Knotting Element for Tissue Closure Post-Endoscopic Mucosal Resection (EMR) Tissue Apposition.
Description: The total number of participants with successful deployments of tissue anchors and associated knotting elements for tissue closure post-Endoscopic Mucosal Resection (EMR) tissue apposition and achieving defect closure.
Time Frame: 3 month follow-up
Measure: Number; unit: participants
Arm/Group | Enrolled Subjects Treated With Tissue Apposition System (TAS)
Number analyzed (Participants) | 7
participants | 6

2. Secondary Outcome: Number of Participants With Durable Tissue Appositions at Three Months Post-Endoscopic Mucosal Resection (EMR) Tissue Apposition
Time Frame: 3 month follow-up
Population: All enrolled subjects were analyzed
Measure: Number; unit: Participants
Arm/Group | Enrolled Subjects Treated With Tissue Apposition System (TAS)
Number analyzed (Participants) | 7
Participants | 6

3. Primary Outcome: Numbers of Participants With Successful Deployment of Tissue Apposition System (TAS)
Description: Number of enrolled subjects (participants) treated with successful deployment of the Tissue Apposition System (TAS) device.
Time Frame: At The Time of Surgery
Population: All enrolled subjects were analyzed
Measure: Number; unit: participants
Arm/Group | Enrolled Subjects Treated With Tissue Apposition System (TAS)
Number analyzed (Participants) | 7
participants | 6

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Enrolled Subjects Treated With Tissue Apposition System (TAS)
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects Treated With Tissue Apposition System (TAS) (N=7)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) — The EMR procedure was performed on 12 March 2008. Two days later, on 14 March 2008, the subject underwent elective spinal surgery for his ongoing stenosis. In the opinion of the PI, this SAE was unrelated to the EMR procedure or TAS.
Chest Pain (Cardiac disorders) | 1 (1) — EMR was performed on 05May2008. On 18May2008, subject had moderate chest pain requiring hospitalization. Following pharmaceutical intervention, resolved without sequelae 3 days after onset. In the opinion of the PI, this SAE was unrelated to TAS.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Subjects Treated With Tissue Apposition System (TAS) (N=7)
Abdominal Pain (General disorders) | 6 (7)
Abdominal Tenderness (General disorders) | 4 (4)
Hypotension (General disorders) | 1 (1)
scratch (Skin and subcutaneous tissue disorders) | 1 (1)
hemoglobin low (Blood and lymphatic system disorders) | 1 (1)
sinus bradycardia (Cardiac disorders) | 1 (1)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 (1)
Abdominal cramp (General disorders) | 3 (4)
blood in stool (Gastrointestinal disorders) | 2 (2)
dry mouth (Skin and subcutaneous tissue disorders) | 1 (1)
headache (Nervous system disorders) | 3 (3)
lower abdominal pain (General disorders) | 1 (1)
numbness lips (Skin and subcutaneous tissue disorders) | 2 (2)
Shoulder discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
tingling lips (Skin and subcutaneous tissue disorders) | 2 (2)
pain abdominal (General disorders) | 1 (1)
granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
pain in toe (Musculoskeletal and connective tissue disorders) | 1 (1)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
application site bruise (Skin and subcutaneous tissue disorders) | 1 (1)
hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 2 (2)
injection site itching (Skin and subcutaneous tissue disorders) | 1 (1)
low hemoglobin (Blood and lymphatic system disorders) | 1 (1)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
abdominal aortic aneurysm (Vascular disorders) | 1 (1)
low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
dry nose (General disorders) | 1 (1)
RBC low (Blood and lymphatic system disorders) | 1 (1)
soreness corner of mouth (General disorders) | 2 (2)
suture line inflammation (Surgical and medical procedures) | 1 (1)
abdominal bloating (Gastrointestinal disorders) | 1 (1)
tenderness (General disorders) | 1 (1)
polyp removal (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days